CLINICAL TRIAL: NCT04209452
Title: Improving Working Memory of Children With Autism Through Instruction on Rehearsal Strategy and Reinforcement
Brief Title: Improving Working Memory of Children With Autism
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Arizona State University (Other)
Collaborators: Shanghai Xuhui Clover Children Healthy Garden (Unknown); Jingdezhen Kindkids Autism Rehabilitation and Training Center (Unknown); Sunshine Special Education Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00010960
Record Dates: First submitted 2019-12-09; First posted 2019-12-24 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Reinforcement Machine Learning

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): No intervention will be provided for participants enrolled in the control group.
- Rehearsal (Experimental): Participants will receive instruction on rehearsal strategy.
  Interventions: Behavioral: Rehearsal strategy
- Reinforcement (Experimental): Participants will receive reinforcement for correct recall.
  Interventions: Behavioral: Reinforcement
- Rehearsal + Reinforcement (Experimental): The participants in this group will receive instruction on rehearsal strategy and reinforcement for correct recall.
  Interventions: Behavioral: Rehearsal strategy and reinforcement

INTERVENTIONS:
Behavioral: Rehearsal strategy — Teaching children to cumulatively rehearse numbers as they are being said.
  Arms: Rehearsal
Behavioral: Reinforcement — Providing reinforcement for correct recall after a delay.
  Arms: Reinforcement
Behavioral: Rehearsal strategy and reinforcement — Teaching children to cumulatively rehearse numbers as they are being said, AND providing reinforcement for correct recall after a delay.
  Arms: Rehearsal + Reinforcement

SUMMARY:
Existing findings suggest that challenges in working memory (WM) of children with autism are common (Habib, Pollick, Melville, & 2019). The WM malfunction can last across the lifespan and individuals with autism exhibit large WM impairments in both phonological and visuospatial domains (Habib, Harris, Pollick & Melville, 2019). Despite the well-documented effects of WM impairments, little research has been dedicated to strategies for improving the working memory of children with autism.

Previous research found that individuals who verbally repeat a previously presented stimulus (i.e., rehearsal) tended to perform better than those who do not rehearse (Bebko, Rhee, Ncube, & Dahary, 2017; Joseph, Steele, Meyer, & Tager-Flusberg, 2005). In addition, among studies that investigated WM in children with autism, Baltruschat et al (2011a; 2011; 2012) conduct studies using positive reinforcement. Their results reveal that the positive reinforcement appeared to have produced better working memory.

The present study intends to investigate if training children with autism to use rehearsal strategy would improve their working memory. In addition, the investigators are also interested to see if reinforcement is a critical component that may provide additive effects beyond the effects of rehearsal. The investigators intend to randomly assign children to four different conditions: control, rehearsal, reinforcement, and rehearsal + reinforcement conditions. The results of this study should provide empirical evidence for practitioners to improve WM in children with autism.

DETAILED DESCRIPTION:
Prescreening:

The purpose of prescreening is to determine the IQ and functioning level of the participants. The investigators will administrate IQ tests in which the participants will complete a series of tasks such as pointing to images/objects, placing objects, and answer questions upon instruction. The investigators will interview parents regarding their children's levels of functioning as well as their information (e.g., level of education). Additionally, the investigators will also assess the number of digits (digit span) and delay for each participant as the participants may function at different levels. Members of the research team will test a combination of different digit span and delays for each participant to assess how many digits in a sequence (i.e., digit span) they can remember and how long (i.e., delay) they can remember the digit sequence.

Pretest:

A pretest trial starts when a teacher asks a participant to repeat a sequence of numbers and a sequence of nonsense words. The teacher will say one number or one nonsense word at a time, wait for a predetermined interval, and ask the participant to report the numbers or the words in the exact sequence as they hear. The trial ends after the participant recalls correctly or incorrectly, or if the participant does not produce a recall after 5 s. The teacher will not provide any verbal feedback for participants' responses during the pretest. The investigators will conduct pretest for approximately one week. During the pretest, teacher will record exactly what the participant says.

Random assignment:

After pretest, the participants will be randomly assigned to one of four groups: control, rehearsal, reinforcement, and rehearsal + reinforcement groups.

Control group Participants in this group will not receive any intervention during the study.

Rehearsal group Participants in this group will receive rehearsal intervention. The intervention will last approximately 2-3 weeks depending on the participant performance. Sessions will be conducted daily, and each will include 10 trials.

A preference assessment will be conducted to determine the reinforcer before each session. Participants will be asked to choose a reinforcer that they would like to receive during the instruction. In a rehearsal trial, the teacher will verbally present numbers in a sequence. After a number is verbally presented, the teacher will prompt the participant to rehearse (repeat) the number being said as well as all previous numbers. Correct rehearsal will be followed by a reinforcer (e.g., an edible item with verbal praise). Once the participant can independently rehearse the number(s), the prompts for verbal rehearsal will only be provided when he or she does not start providing a rehearsal within 1 s. The reinforcer will then only be given for correct unprompted verbal rehearsal. If the participant does not provide any verbal rehearsals or verbalize incorrect numbers, the instructor will repeat the process and ask the participant to rehearse the numbers again. After the predetermined delay after the correct verbal rehearsal, the participant will be asked to recall the number sequence. No reinforcement or feedback will be provided.

Reinforcement group A preference assessment will be conducted to determine the reinforcer before each session. Participants will be asked to choose a reinforcer that they would like to receive during the instruction. Before each trial, the teacher will verbally instruct the participant to try to remember the numbers and that the reinforcer will be delivered upon the correct recall. In each trial, the teacher will verbally present numbers in a sequence. After a while, the teacher will ask the participant to repeat the numbers in the sequence. If the participant correctly repeats the numbers, the reinforcer will be given. If the numbers are repeated incorrectly, the reinforcement will not be given. No other instruction will be given (e.g., on rehearsal strategy).

Rehearsal + reinforcement group The participants in this group will receive rehearsal intervention and reinforcement in the same manner as the participants in the rehearsal group as well as in the reinforcement group.

Posttest:

Posttest procedure and data collection will be the same as those during pretest.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of autism
* have an echoic repertoire

Exclusion Criteria:

* problem behavior or noncompliance

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2020-11-10 (Actual)

PRIMARY OUTCOMES:
Change in percent recall | Before, during, and up to 2 weeks after intervention.
  Participants will hear a sequence of digits or words (range from 1 to 9 stimuli) and then will be asked to recall the serial order after a delay (e.g., 9, 12, or 15 s). Percent correct recall of serial order will be calculated for all sequences as well as for each sequence size and delay. Change of percent recall from before, during, and after the intervention will be measured.

SECONDARY OUTCOMES:
Change in percent strategy used. | During the intervention, and up to 2 weeks after intervention.
  Percentage of trials in which a rehearsal strategy or another memory strategy is used will be calculated during and after the intervention. We will code the strategies used by participants and calculate the percentage of trials in which a rehearsal strategy or another strategy they used.

CONTACTS AND LOCATIONS:
Overall Officials: Chengan Yuan, PhD, Principal Investigator — Arizona State University; Erin Rotheram-Fuller, PhD, Principal Investigator — Arizona State University
Locations (3):
- China (3):
  - Jingdezhen Kindkids Autism Rehabilitation and Training Center, Jingdezhen, Jiangxi
  - Sunshine Special Education Center, Taizhou, Zhejiang
  - Shanghai Xuhui Clover Children Healthy Garden, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Habib A, Harris L, Pollick F, Melville C. A meta-analysis of working memory in individuals with autism spectrum disorders. PLoS One. 2019 Apr 30;14(4):e0216198. doi: 10.1371/journal.pone.0216198. eCollection 2019. PMID 31039192
- [Background] Joseph RM, Steele SD, Meyer E, Tager-Flusberg H. Self-ordered pointing in children with autism: failure to use verbal mediation in the service of working memory? Neuropsychologia. 2005;43(10):1400-11. doi: 10.1016/j.neuropsychologia.2005.01.010. Epub 2005 Feb 17. PMID 15989932
- [Background] Baltruschat L, Hasselhorn M, Tarbox J, Dixon D R, Najdowski AC, Mullins R D, Gould, ER. Addressing working memory in children with autism through behavioral intervention. Research in Autism Spectrum Disorders. 2011;5(1): 267-76. doi: 10.1016/j.rasd.2010.04.008
- [Background] Bebko JM, Rhee T, Ncube BL, Dahary H. Effectiveness and Retention of Teaching Memory Strategy Use to Children With Autism Spectrum Disorder. Canadian Journal of School Psychology. 2017;32(3-4): 244-64. doi: 10.1177/0829573517699332